CLINICAL TRIAL: NCT03711929
Title: LUMINA: A Phase III, Multicenter, Sham-Controlled, Randomized, Double-Masked Study Assessing the Efficacy and Safety of Intravitreal Injections of 440 ug DE-109 for the Treatment of Active, Non-Infectious Uveitis of the Posterior Segment of the Eye.
Brief Title: LUMINA Phase III Study Assessing the Efficacy and Safety of Intravitreal Injections of 440 ug DE-109 Sirolimus for the Treatment of Active, Non-Infectious Uveitis of the Posterior Segment of the Eye
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business decision
Sponsor: Santen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 010906IN
Record Dates: First submitted 2018-10-17; First posted 2018-10-19 (Actual); Results first posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Non Infectious Uveitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Test Arm: DE-109 Injectable Solution (Experimental): Intravitreal injection of DE-109 440 µg in the study eye(s) every 2 months (Day 1, Month 2, and Month 4).
  Interventions: Drug: DE-109 Intravitreal Injections
- Control Arm: Sham Procedure (Sham Comparator): Sham procedure administered to the study eye(s) every 2 months (Day 1, Month 2, and Month 4). The sham procedure mimics an intravitreal injection without penetrating the eye.
  Interventions: Other: Sham Procedure
- Dummy Arm: DE-109 Injectable Solution (Other): Dummy Arm: Intravitreal injection of DE-109 at an undisclosed, fixed dose (within the range of 44 µg to 880 µg) in the study eye(s) every 2 months (Day 1, Month 2, and Month 4).
  Interventions: Drug: DE-109 Intravitreal Injections
- Open-label:DE-109 Injectable Solution (Experimental): Subjects completing the Month 6 pre-dose evaluations (the final evaluations in the double-masked period) began the open-label period of the study, in which all subjects received intravitreal injection of DE-109 440 μg in the study eye(s) every 2 months for an additional 6 months of dosing.
  Interventions: Drug: DE-109 Intravitreal Injections (Open Label)

INTERVENTIONS:
Drug: DE-109 Intravitreal Injections — 440 ug of DE-109 Injectable Solution
  Arms: Test Arm: DE-109 Injectable Solution
Other: Sham Procedure — The sham procedure mimics an intravitreal injection without penetrating the eye.
  Arms: Control Arm: Sham Procedure
Drug: DE-109 Intravitreal Injections — Undisclosed Fixed Dose of DE-109 Injectable Solution (range of 44 ug to 880 ug)
  Arms: Dummy Arm: DE-109 Injectable Solution
Drug: DE-109 Intravitreal Injections (Open Label) — After double-masked treatment period (injections every 2 months), eligible subjects would enter the open-labeled period and had DE-109 440 ug injections every 2 months (Month 6, Month 8, and Month 10)
  Arms: Open-label:DE-109 Injectable Solution

SUMMARY:
This is a Phase III study to assess the efficacy and safety of DE-109 440 µg every 2 months in subjects with active, non-infectious uveitis of the posterior segment of the eye (NIU-PS).

There is a 6-month, single-arm, open-label period after completion of the 6-month double- masked, controlled period allows the evaluation of the efficacy and safety of intravitreal injection of DE-109 440 µg every 2 months for longer duration than appropriate for a placebo or sham control.

ELIGIBILITY:
Inclusion Criteria:

Non-Infectious Active Uveitis of the Posterior Segment

Exclusion Criteria:

Females who are pregnant, nursing, or planning a pregnancy Confirmed or suspected infectious uveitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2022-06-14 (Actual); Study Completion 2022-06-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (65):
- United States (38):
  - Arizona Retina & Vitreous Consultants, Phoenix, Arizona
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Kaiser Permanente Medical Center, Los Angeles, California
  - USC Roski Eye Institute, Los Angeles, California
  - Byers Eye Institute at Stanford, Palo Alto, California
  - California Eye Specialist Medical Group, Inc., Pasadena, California
  - Colorado Retina Associates, Golden, Colorado
  - Retina Vitreous Associates of Florida, St. Petersburg, Florida
  - University of South Florida Eye Institute, Tampa, Florida
  - Emory Eye Center, Atlanta, Georgia
  - Marietta Eye Clinic, Marietta, Georgia
  - Cook County Health & Hospitals System, Chicago, Illinois
  - Illinois Retina Associate, Oak Park, Illinois
  - Raj K.Maturi, MD, Indianapolis, Indiana
  - University of Kansas School of Medicine, Prairie Village, Kansas
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Kresge Eye Institute, Detroit, Michigan
  - Associated Retina Consultants-Royal Oak, Royal Oak, Michigan
  - Discover Vision Center, Independence, Missouri
  - Eye Associates of New Mexico, Albuquerque, New Mexico
  - New York Eye & Ear Infirmary of Mt. Sinai, New York, New York
  - Wake Forest Baptist Medical Center/Surgery, Winston-Salem, North Carolina
  - Cleveland Clinic Cole Eye Institute, Cleveland, Ohio
  - Cascade Medical Research Institute, LLC, Eugene, Oregon
  - Retina Vitreous Consultants, Monroeville, Pennsylvania
  - Mid Atlantic Retina, Philadelphia, Pennsylvania
  - UPMC Eye Center, Pittsburgh, Pennsylvania
  - Vanderbilt Eye Institute, Nashville, Tennessee
  - Austin Retina Associate, Austin, Texas
  - Texas Retina Associates-Dallas-Main, Dallas, Texas
  - Houston Eye Associates, Houston, Texas
  - Retina Consultants of Houston, Houston, Texas
  - Valley Retina Institute, McAllen, Texas
  - Foresight Studies, San Antonio, San Antonio, Texas
  - Medical Center Ophthalmology Associate, San Antonio, Texas
  - Retina Group of Washington, Fairfax, Virginia
  - West Virginia University Eye Institute, Morgantown, West Virginia
- Argentina (8):
  - Centro De Ojos Loria SRL, Lomas de Zamora, Buenos Aires
  - Clinica Privada de Ojos, Mar del Plata, Buenos Aires
  - Primer Hospital Privado De Ojos, Buenos Aires, Buenos Aires F.D.
  - Hospital Universitario Austral, Buenos Aires, Buenos Aires F.D.
  - Gustavo Ariel Budmann Private Office, Buenos Aires, Odisha
  - Oftalmologia Global, Rosario, Santa Fe Province
  - Organización Médica de Investigación (OMI), Caba
  - Centro Privado de Ojos Romagosa Fundacion VER, Córdoba
- India (14):
  - Sri Sankaradeva Nethralaya, Guwahati, Assam
  - Banker's Retina Clinic & Laser Centre, Ahmedabad, Gujarat
  - Narayana Nethralaya, Bangalore, Karnataka
  - Disha Eye Hospitals Pvt Ltd, Pune, Maharashtra
  - PBMA'S H. V. Desai Eye Hospital, Pune, Maharashtra
  - LV Prasad Eye Institute, Bhubaneswar, Odisha
  - SMS Hospital, Jaipur, Rajasthan
  - Sankara Nethralaya, Chennai, Tamil Nadu
  - Aravind Eye Hospital (Coimbatore), Coimbatore, Tamil Nadu
  - Aravind Eye Hospitals, Madurai, Tamil Nadu
  - L V Prasad Eye Institute, Hyderabad, Telangana
  - Dr. J.L. Rohatgi Memorial Eye Hospital, Kanpur, Uttar Pradesh
  - BB Eye Foundation, Kolkata, West Bengal
  - Advanced Eye Center, Chandigarh
- Italy (5):
  - Polo Universita degli Studi di Milano Ospedale Luigi Sacco Clinca Oculistica (Eye Clinic), Milan, Lombardy
  - Universita degli Studi di Padova - Azienda Ospedaliera di Padova - Clinica Oculistica, Padua, Veneto
  - A.O.U. Policlinico SantOrsola-Malpigi, Bologna
  - San Raffaele Scientific Institute, Milan
  - Azienda USL IRCCS Reggio Emilia, Reggio Emilia

REFERENCES:
- [Derived] Hashida N, Nishida K. Recent advances and future prospects: Current status and challenges of the intraocular injection of drugs for vitreoretinal diseases. Adv Drug Deliv Rev. 2023 Jul;198:114870. doi: 10.1016/j.addr.2023.114870. Epub 2023 May 10. PMID 37172783

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Study Eyes
Groups:
- Dummy Arm: DE-109 Injectable Solution: Dummy Arm: Intravitreal injection of DE-109 at an undisclosed, fixed dose (within the range of 44 µg to 880 µg) in the study eye(s) every 2 months (Day 1, Month 2, and Month 4). This study arm has the same route of administration and frequency as the test arm.
  DE-109 Intravitreal Injections: Undisclosed Fixed Dose of DE-109 Injectable Solution (range of 44 ug to 880 ug).
Period: Double Masked Treatment Period (DMTP)
Arm/Group | Test Arm: DE-109 Injectable Solution | Control Arm: Sham Procedure | Dummy Arm: DE-109 Injectable Solution
Started | 57; 65 Study Eyes (Units assigned to Arm/Group are whole participants. If participants enrolled both eyes to the study, both eyes received the same assigned intervention.) | 59; 68 Study Eyes (Units assigned to Arm/Group are whole participants. If participants enrolled both eyes to the study, both eyes received the same assigned intervention.) | 29; 32 Study Eyes (Units assigned to Arm/Group are whole participants. If participants enrolled both eyes to the study, both eyes received the same assigned intervention.)
Completed | 51; 59 Study Eyes (Units assigned to Arm/Group are whole participants. If participants enrolled both eyes to the study, both eyes received the same assigned intervention.) | 48; 55 Study Eyes (Units assigned to Arm/Group are whole participants. If participants enrolled both eyes to the study, both eyes received the same assigned intervention.) | 24; 27 Study Eyes (Units assigned to Arm/Group are whole participants. If participants enrolled both eyes to the study, both eyes received the same assigned intervention.)
Not Completed | 6; 6 Study Eyes | 11; 13 Study Eyes | 5; 5 Study Eyes
Period: Open Label Treatment Period (OLTP)
Arm/Group | Test Arm: DE-109 Injectable Solution | Control Arm: Sham Procedure | Dummy Arm: DE-109 Injectable Solution
Started | 42; 49 Study Eyes (Some participants exited the study or got rescued during Double Masked Treatment Period, hence, less participants entered the Open Label Treatment Period in the Test arm. Units assigned to Arm/Group are whole participants. If participants enrolled both eyes to the study, both eyes received the same assigned intervention.) | 40; 47 Study Eyes (Some participants exited the study or got rescued during Double Masked Treatment Period, hence, less participants entered the Open Label Treatment Period in the Control arm. Units assigned to Arm/Group are whole participants. If participants enrolled both eyes to the study, both eyes received the same assigned intervention.) | 21; 24 Study Eyes (Some participants exited the study or got rescued during Double Masked Treatment Period, hence, less participants entered the Open Label Treatment Period in the Dummy arm. Units assigned to Arm/Group are whole participants. If participants enrolled both eyes to the study, both eyes received the same assigned intervention.)
Completed | 34; 40 Study Eyes (Units assigned to Arm/Group are whole participants. If participants enrolled both eyes to the study, both eyes received the same assigned intervention.) | 35; 41 Study Eyes (Units assigned to Arm/Group are whole participants. If participants enrolled both eyes to the study, both eyes received the same assigned intervention.) | 15; 16 Study Eyes (Units assigned to Arm/Group are whole participants. If participants enrolled both eyes to the study, both eyes received the same assigned intervention.)
Not Completed | 8; 9 Study Eyes | 5; 6 Study Eyes | 6; 8 Study Eyes

BASELINE CHARACTERISTICS:
Groups:
- Dummy Arm: DE-109 Injectable Solution: Dummy Arm: Intravitreal injection of DE-109 at an undisclosed, fixed dose (within the range of 44 µg to 880 µg) in the study eye(s) every 2 months (Day 1, Month 2, and Month 4). This study arm (which has the same route of administration and frequency as the test arm).
  DE-109 Intravitreal Injections: Undisclosed Fixed Dose of DE-109 Injectable Solution (range of 44 ug to 880 ug)
- Total: Total of all reporting groups
Arm/Group | Test Arm: DE-109 Injectable Solution | Control Arm: Sham Procedure | Dummy Arm: DE-109 Injectable Solution | Total
Number analyzed (Participants) | 57 | 59 | 29 | 145
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (17.26) | 46.2 (14.40) | 47.0 (14.27) | 46.6 (15.46)
Age, Customized [Count of Participants; unit: Participants]
  <65 | 47 | 52 | 27 | 126
  >= 65 years | 10 | 7 | 2 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 35 | 14 | 85
  Male | 21 | 24 | 15 | 60
Race (NIH/OMB) [Count of Participants; unit: Participants] — The sum of the participants in the "total" Arm/Group is 145 and is consistent with the overall number of Baseline Participants of 145.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 19 | 18 | 11 | 48
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
    Black or African American | 8 | 7 | 6 | 21
    White | 29 | 33 | 12 | 74
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Argentina | 12 | 9 | 3 | 24
  United States | 26 | 31 | 14 | 71
  Italy | 1 | 3 | 1 | 5
  India | 18 | 16 | 11 | 45

OUTCOME MEASURES:

1. Primary Outcome: Vitreous Haze (VH) of Zero Response at Month 5
Description: Vitreous Haze (VH) was assessed during slit-lamp biomicroscopy and scored using the modified Standardized Uveitis Nomenclature (SUN) scale as follows:
  * Score = 0: No inflammation
  * Score = 0.5+: Trace inflammation (slight blurring if the optic disc margins and/or loss of nerve fiber layer reflex)
  * Score = 1+: Mild blurring of the retinal vessels and optic nerve
  * Score = 1.5+: Optic nerve had and posterior retina view obstruction greater than 1+ but less than 2+
  * Score = 2+: Moderate blurring of the optic nerve head
  * Score = 3+: Marked blurring of the optic nerve head
  * Score = 4+: Optic nerve head not visible
  VH 0 response (resolution of inflammation) is defined as a VH score of 0 in the study eye at a specified follow up visit based on the modified SUN scale.
  The response as a percentage is calculated as the proportion of study eyes which achieved a VH score of zero at Month 5
Time Frame: Month 5
Population: Full Analysis Set
Measure: Number; unit: percentage response of study eyes
Units Other Than Participants: Study Eyes
Arm/Group | Test Arm: DE-109 Injectable Solution | Control Arm: Sham Procedure | Dummy Arm: DE-109 Injectable Solution
Number analyzed (Participants) | 57 | 59 | 29
Number analyzed (Study Eyes) | 65 | 68 | 32
percentage response of study eyes | 15.7 | 12.2 | 28.7

2. Secondary Outcome: Mean Composite Score at Month 3 and Month 5
Description: Composite score scale is defined as follows. Each study eye was assigned one of the following scores:
  * Score = 3 if a study eye achieved Vitreous Haze (VH) score of 0 at the specified visit without taking any rescue therapies that could affect VH score prior to the specified visit.
  * Score = 2 if a study eye had at least improved (decreased) by 2 units (i.e., 2+ to 0, 3+ to 1+, or 4+ to 2+) in VH (compared to baseline) at the specified visit without taking any rescue therapies that could affect VH score prior to the specified visit.
  * Score = 1 if a study eye achieved VH score of 0.5+ at the specified visit without taking any rescue therapies that could affect VH score prior to the specified visit.
  * Score = -1 if a study eye got rescued due to worsening of uveitis or discontinued from the study due to lack of efficacy or due to adverse event prior to the specified visit.
  * Score = 0 if otherwise
Time Frame: Month 3, Month 5
Population: Full Analysis Set. The number of overall participants analyzed is consistent with data here and other parts of the record. Data represented in all records are for whole participants. Subjects with two study eyes had the composite score as the average score of both eyes.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Test Arm: DE-109 Injectable Solution | Control Arm: Sham Procedure | Dummy Arm: DE-109 Injectable Solution
Number analyzed (Participants) | 57 | 59 | 29
score on a scale
  Month 3 | 0.4 (1.10) | 0.3 (0.80) | 0.4 (0.98)
  Month 5 | 0.3 (1.11) | 0.3 (1.04) | 0.6 (1.31)

3. Secondary Outcome: Vitreous Haze (VH) of Zero Response at Month 3
Description: Vitreous Haze (VH) was assessed during slit-lamp biomicroscopy and scored using the modified Standardized Uveitis Nomenclature (SUN) scale as follows:
  * Score = 0: No inflammation
  * Score = 0.5+: Trace inflammation (slight blurring if the optic disc margins and/or loss of nerve fiber layer reflex)
  * Score = 1+: Mild blurring of the retinal vessels and optic nerve
  * Score = 1.5+: Optic nerve had and posterior retina view obstruction greater than 1+ but less than 2+
  * Score = 2+: Moderate blurring of the optic nerve head
  * Score = 3+: Marked blurring of the optic nerve head
  * Score = 4+: Optic nerve head not visible
  VH 0 response (resolution of inflammation) is defined as a VH score of 0 in the study eye at a specified follow up visit based on the modified SUN scale.
  The response as a percentage is calculated as the proportion of study eyes which achieved a VH score of zero at Month 3.
Time Frame: Month 3
Population: Full Analysis Set
Measure: Number; unit: percentage response of study eyes
Units Other Than Participants: Study Eyes
Arm/Group | Test Arm: DE-109 Injectable Solution | Control Arm: Sham Procedure | Dummy Arm: DE-109 Injectable Solution
Number analyzed (Participants) | 57 | 59 | 29
Number analyzed (Study Eyes) | 65 | 68 | 32
percentage response of study eyes | 14.7 | 5.5 | 15.4

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent and were followed to resolution or until the subject's participation in the study ended for both periods: 6-month Double-Masked Treatment Period at Month 6; and 6-month Open-Label Treatment Period at Month 12.
Groups:
- DE-109 440 μg (Double Masked Treatment Period): Intravitreal injection of DE-109 440 µg in the study eye(s) every 2 months (Day 1, Month 2, and Month 4).
  DE-109 Intravitreal Injections: 440 ug of DE-109 Injectable Solution
- Sham Procedure (Double Masked Treatment Period): Sham procedure administered to the study eye(s) every 2 months (Day 1, Month 2, and Month 4). The sham procedure mimics an intravitreal injection without penetrating the eye.
  Sham Procedure: The sham procedure mimics an intravitreal injection without penetrating the eye.
- DE-109 Fixed Dose (Double Masked Treatment Period): Dummy Arm: Intravitreal injection of DE-109 at an undisclosed, fixed dose (within the range of 44 µg to 880 µg) in the study eye(s) every 2 months (Day 1, Month 2, and Month 4). This study arm has the same route of administration and frequency as the test arm).
  DE-109 Intravitreal Injections: Undisclosed Fixed Dose of DE-109 Injectable Solution (range of 44 ug to 880 ug)
- DE-109 440 μg/DE-109 440 μg (Open Label Treatment Period); Sham/DE-109 440 μg (Open Label Treatment Period); DE-109 Fixed Dose/DE-109 440 μg (Open Label Treatment Period): a 6-month open-label period in which all subjects continued to receive DE 109 440 μg every 2 months in the study eye.
Arm/Group | DE-109 440 μg (Double Masked Treatment Period) | Sham Procedure (Double Masked Treatment Period) | DE-109 Fixed Dose (Double Masked Treatment Period) | DE-109 440 μg/DE-109 440 μg (Open Label Treatment Period) | Sham/DE-109 440 μg (Open Label Treatment Period) | DE-109 Fixed Dose/DE-109 440 μg (Open Label Treatment Period)
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/59 | 0/29 | 0/42 | 0/40 | 0/21
Serious Adverse Events (participants affected / at risk) | 7/57 | 3/59 | 5/29 | 3/42 | 1/40 | 0/21
Other Adverse Events (participants affected / at risk) | 47/57 | 45/59 | 22/29 | 31/42 | 25/40 | 8/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DE-109 440 μg (Double Masked Treatment Period) (N=57) | Sham Procedure (Double Masked Treatment Period) (N=59) | DE-109 Fixed Dose (Double Masked Treatment Period) (N=29) | DE-109 440 μg/DE-109 440 μg (Open Label Treatment Period) (N=42) | Sham/DE-109 440 μg (Open Label Treatment Period) (N=40) | DE-109 Fixed Dose/DE-109 440 μg (Open Label Treatment Period) (N=21)
Uveitis (Eye disorders) | 2 | 0 | 1 | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 2 | 0 | 0 | 0
Angle closure glaucoma (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Birdshot chorioretinopathy (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Blindness (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Iridocyclitis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Non-infectious endophthalmitis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Endophthalmitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Chorioretinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Eye abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Brain injury (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Strangulated hernia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Toxic anterior segment syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DE-109 440 μg (Double Masked Treatment Period) (N=57) | Sham Procedure (Double Masked Treatment Period) (N=59) | DE-109 Fixed Dose (Double Masked Treatment Period) (N=29) | DE-109 440 μg/DE-109 440 μg (Open Label Treatment Period) (N=42) | Sham/DE-109 440 μg (Open Label Treatment Period) (N=40) | DE-109 Fixed Dose/DE-109 440 μg (Open Label Treatment Period) (N=21)
Uveitis (Eye disorders) | 9 | 12 | 5 | 5 | 4 | 2
Cystoid macular oedema (Eye disorders) | 6 | 11 | 1 | 3 | 4 | 0
Conjunctival haemorrhage (Eye disorders) | 7 | 5 | 4 | 6 | 4 | 1
Iridocyclitis (Eye disorders) | 7 | 4 | 3 | 2 | 2 | 1
Cataract (Eye disorders) | 4 | 1 | 4 | 4 | 3 | 0
Cataract subcapsular (Eye disorders) | 3 | 3 | 3 | 2 | 1 | 0
Eye pain (Eye disorders) | 4 | 1 | 1 | 0 | 2 | 1
Macular oedema (Eye disorders) | 1 | 4 | 1 | 0 | 1 | 0
Ocular hyperaemia (Eye disorders) | 4 | 0 | 1 | 0 | 1 | 0
Vitreous floaters (Eye disorders) | 0 | 3 | 0 | 0 | 4 | 1
Iris adhesions (Eye disorders) | 2 | 1 | 2 | 1 | 2 | 0
Visual impairment (Eye disorders) | 3 | 0 | 1 | 3 | 0 | 0
Eye irritation (Eye disorders) | 1 | 0 | 2 | 0 | 1 | 0
Keratic precipitates (Eye disorders) | 0 | 2 | 2 | 1 | 1 | 0
Intraocular pressure increased (Investigations) | 15 | 8 | 3 | 9 | 8 | 1
Product residue present (Investigations) | 4 | 1 | 4 | 1 | 2 | 1
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 2 | 0 | 0 | 0
Chorioretinitis (Infections and infestations) | 1 | 5 | 1 | 1 | 2 | 0
Headache (Nervous system disorders) | 3 | 1 | 1 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-07-14): https://cdn.clinicaltrials.gov/large-docs/29/NCT03711929/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-16): https://cdn.clinicaltrials.gov/large-docs/29/NCT03711929/SAP_001.pdf